CLINICAL TRIAL: NCT01002716
Title: Cell Immunity Response to Vaccination Against Influenza in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Ori Elkayam, Tel Aviv Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TASMC-09-OE-0453-CTIL
Record Dates: First submitted 2009-10-15; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid influenza vaccine cell immunity
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Agrippal S1 (Influenza vaccination) — Single dose of vaccine
  Other Names: Agripal S1

SUMMARY:
The efficacy of vaccination against influenza in patients with rheumatoid arthritis has been assessed using humoral response. However, the cellular immunity is another important pathway of response to vaccination. The purpose of this study is to evaluate the degree of cellular immunity response to influenza vaccination. Patient with rheumatoid arthritis and healthy controls will participate in this study , will undergo a clinical evaluation the day of vaccination and 4 weeks after. The humoral and cell immunity response will be assessed the day of vaccination and 4 weeks later

DETAILED DESCRIPTION:
Sixty patients with RA and 30 healthy , aged matched controls will participate in the study.

After signing informed consent, all subjects will be vaccinated with the inactivated split virion vaccine which will be recommended by the WHO next fall.

Patients will be evaluated at weel 0 and 6 weeks later. Clinical evaluation will be based on the Disease Activity Score 28 (DAS 28) which includes number of swollen and tender joints, visual global evaluation of the physician , ESR and CRP Blood with be collected on the day of vaccination and 6 weeks later.

Preparation of peripheral blood mononuclear cells Blood samples will be obtained prior to and 4 weeks after vaccination. Peripheral blood mononuclear cells (PBMC) will be isolated by centrifugation of heparinized blood on a Lymphoprep gradient (Nycomed, Oslo, Norway). Cells will be washed twice in tissue culture medium RPMI (RPMI1640-Hepes with Glutamax-I, GIBCO BRL, NY, USA) and resuspended to a concentration of 2 106/ml in RPMI 1640 supplemented with 10% heat inactivated fetal bovine serum (FBS) (GIBCO BRL, NY, USA).

ELISPOT assay The 96-well PVDF (polyvinylidene difluoride, Millipore Corp., MA, USA) plates will be prewet with 70% EtOH, then coated with 100 l/well of anti-human IFN- monoclonal antibody (mAb) 1-D1K , diluted to 15 g/ml in sterile filtered phosphate-buffered saline (PBS) . The plates will be kept overnight at 4°C. A total of 100 000 PBMC plus 5 l/well (1 g/ml) peptides will be added to each well in duplicate for each condition and incubated for 24 h at 37°C in 5% CO2. After incubation the plates will be washed with PBS then 100 l of biotinylated mAb (7-B6-1-biotin, Mabtech AB), diluted in filtered PBS with 0.5% FBS to the concentration 1 g/ml were added to each well. The plates will be incubated 2 h at room temperature, washed with PBS and then incubated with 100 l/well of streptavidine-alkaline phosphatase (Mabtech AB) diluted 1-1000 in PBS with 0.5% FBS for 1 h at room temperature. After washing, cells will be developed by adding 100 l/well of colorimetric substrate (BCIP/NBT-plus, Mabtech AB) and then counted in an ELISPOT reader. Each spot was produced by a single IFN- secreting T-cell-spot-forming cell (SFC). All tests were performed in duplicate and the mean values were calculated. A response will be considered to be positive when the number of spots in the wells with peptide-stimulated cells, after subtraction of the background (wells without peptide stimulation), will be at least two-fold greater than the number of background spots14 and more than 20/106 SFC.

Detection of intracellular cytokine production by flow cytometry The intracellular staining method will be used for identifying the phenotype of INF- producing T cells activated by peptide stimulation. The staining will be performed using the protocol described by Rauser et al.15 PBMC were stimulated for 6 h with 1 g/ml influenza peptides. Brefeldin A (10 g/ml, Sigma-Aldrich, St Louis, MO) will be added for the last 4 h of the incubation. A positive control will be obtained by stimulating the cells with 0.5 g/ml PMA (Phorbol 12-myrestate 13-acetate) and 1 g/ml Ionomycin (both from Sigma-Aldrich, St Louis, MO, USA). The cells will be permeabilized and stained with fluorochrome-labeled anti-CD3, anti-CD4 or anti-CD8 and anti-IFN- antibodies (Becton Dickinson, San Jose, CA, USA). Samples will be analyzed by flow cytometry using FACSCalibur (Becton Dickinson). The positive limit for this test was 0.05% of IFN producing T cells.

Proliferation of specific CD4+ and CD8+ Cellular response will be evaluated by simultaneously analyzing proliferation of specific T CD4+ and CD8+ lymphocytes upon stimulation with antigens of the three virus strains present in the vaccine and production of activation Th1 cytokines by the same cells.

Briefly, to simultaneously analyze proliferation and cytokine production by influenza specific T cells, peripheral blood mononuclear cells will be obtained at T0 and T1 from each donor, stained with the fluorescent nuclear dye carboxyfluorescein succinimidyl ester (CFSE; Molecular Probes) and cultured in duplicate in the presence of peptides of HA from each of the virus strains contained in the influenza virus vaccine used in the study or control peptide for 72 h. At the end of incubation cultures will be stopped with brefeldin, cells resuspended, stained with fluorochrome-conjugated anti-CD8 and anti-interferon-γ (IFN-γ) monoclonal antibodies (Becton&Dickinson) and analyzed by mean of a six colour flow-cytometer (FACSCanto-Becton&Dickinson) and FACS DIVA software . As at every cell division the nuclear fluorescence is halved, proliferating cells fall in the left quadrants of the cytogram, the more divisions the less fluorescence. IFN-γ producing cells fall in the upper quadrants of the cytograms. Cells that upon specific influenza peptide or control peptide stimulation both proliferate and actively produce IFN-γ (Th1 cytokine) fall in the upper left quadrant of the cytogram. They were measured as frequency (proliferating and IFN-γ-producing cells/total T CD4+ or CD8+ lymphocytes).

Haemagglutination inhibition test The immunogenicity of the vaccine was tested by Haemagglutination inhibition (HI) test.

Influenza virus has two important surface glycoproteins: the haemagglutinin (HA) and the neuraminidase (NA). Antigenic classification and subtyping of influenza viruses is based on these two glycoproteins. HA plays a key role in virus cell entry by binding to cell surface receptors, which are found also on red blood cells of certain species. Binding to red cells results in haemagglutination, which can be observed as a carpet of agglutinated red cells at the bottom of a tube or microtitre well. In the HI test, antibody directed against the viral haemagglutinins block the virus from binding to the blood cells and thus inhibits the haemagglutination reaction.

The pre- and post immunization HI antibodies were tested at the Central Virology Laboratory of the Israeli Ministry of Health using the HI test according to a standard WHO procedure 16. Sera were separated, code labeled, and stored at -20°C until tested. Sera were treated with receptor destroying enzyme cholera filtrate to remove non-specific inhibitors, and with Turkey red blood cells to remove non-specific agglutinins. The treated sera were tested by HI test against the three antigens included in the vaccine: A/California (CAL), B/Shangai (SHAN) and A/New Caledonia (NC). The working dilution (test dose) of each antigen contained four haemagglutinin units in 25 µl of antigen. Test doses were diluted in phosphate buffered saline (PBS) and added to serial dilution of antiserum. The haemagglutinin inhibition titer was determined as the highest dilution of serum that completely inhibits haemagglutination of red blood cells.

The titer of an antiserum not showing any inhibition was recorded as <10. Humoral response was defined as either a fourfold or more rise in titer, or a rise from a non-protective baseline level of <1/40 to 1/40 in HI antibodies four weeks after vaccination 17,18. Geometric mean titers of antibody were calculated to assess the immunity of the whole group.

Primary Endpoint of the study : the proportion of cells producing Interferon gamma in Patients with rheumatoid arthritis and controls Secondary Endpoint: Safety of the vaccine

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis

Exclusion Criteria:

* Allergy to egg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Cell immunity response | 4 weeks

SECONDARY OUTCOMES:
Safety of influenza vaccination | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

REFERENCES:
- See also: Tel Aviv Medical Center — http://www.tasmc.org.il/